CLINICAL TRIAL: NCT04947891
Title: The Establishment of the Integration of Posterior Approach Surgical Treatment and Postoperative Intensive Recovery Management of Patients With Degenerative Cervical Spine Myelopathy
Brief Title: The Establishment of the Integration of Surgery and Postoperative Intensive Recovery of Patients With CSM
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017310
Record Dates: First submitted 2021-06-27; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Cervical Myelopathy; Ossification of Posterior Longitudinal Ligament in Cervical Region
Keywords: Cervical myelopathy; Ossification of posterior longitudinal ligament; Intensive recovery; Quality of life; Surgical outcomes
MeSH Terms: conditions — Ossification of Posterior Longitudinal Ligament

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients will be treated with intensive recovery method after surgery.
  Interventions: Procedure: Intensive recovery management
- Control group: Patients will be treated with regular recovery method after surgery.

INTERVENTIONS:
Procedure: Intensive recovery management — Intensive recovery management includes 3 parts: (1) Preoperative analgesia and airway evaluation. (2) The protection and reconstruction of the musculo-ligamentous complex during the surgery, the safe intubation, and the local infiltration anesthesia during surgery. (3) Collar free, multimodal analgesia, airway management, and early recovery after surgery.
  Groups: Study group

SUMMARY:
This study aims to establish the specialist consensus of the integration of posterior approach surgical treatment and postoperative intensive recovery management for CSM or OPLL patients, and verify its safety, practicability and reliability.

DETAILED DESCRIPTION:
In order to establish the specialist consensus of the integration of posterior approach surgical treatment and postoperative intensive recovery management, and verify its safety, practicability and reliability, this study enrolled 130 patients with CSM or OPLL undergoing C3-7 open-door laminoplasty. Patients are divided in two groups randomly. The study group has 80 patients, treated with postoperative intensive recovery management, and the control group has 50 patients. The data is collected preoperatively, at 3-month follow-up and 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age: 18~70 years. (2) Diagnosed as CSM or OPLL. (3) Going to receive C3-C7 open-door laminoplasty. (4) Agree to join this study and sign the informed consent.

Exclusion Criteria:

* (1) Anterior and posterior combined surgery. (2) Posterior laminoplasty combined fusion. (3) Severe osteoporosis. (4) Morbid obesity. (5) patients with mental disorder. (6) patients with previous history of cervical spine surgery. (7) Abnormal laboratory report of liver function, kidney function and hematologic system.(8) Poor compliance. (9) Patients with other surgical contraindications. (10) Patients with intemperance or taking drugs. (11) Patients who joined other study within the last 3 months.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with degenerative CSM or OPLL undergoing C3-7 open-door laminoplasty
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Cervical spine mechanical analysis | Preoperation to 1 year after surgery.
  The ROM and multi-dimensional mechanical analysis of cervical spine before surgery, at 3-month postoperative follow-up and 1-year follow
Cervical spine functions | Preoperation to 1 year after surgery.
  NDI score and JOACMEQ score before surgery, at 3-month postoperative follow-up and 1-year follow

SECONDARY OUTCOMES:
Outcome of quality of life | Preoperation to 1 year after surgery.
  EQ-5D score before surgery, at 3-month postoperative follow-up and 1-year follow
Outcome of pain | Preoperation to 1 year after surgery.
  VAS score before surgery, at 3-month postoperative follow-up and 1-year follow
Neurological outcome | Preoperation to 1 year after surgery.
  mJOA score before surgery, at 3-month postoperative follow-up and 1-year follow

CONTACTS AND LOCATIONS:
Overall Officials: Feifei Zhou, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Feifei Zhou, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No